CLINICAL TRIAL: NCT05250817
Title: Preferences for the First-Line Treatment of Advanced/Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Preferences for the First-Line Treatment of Advanced/Metastatic Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-69K
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Preference; Advanced/Metastatic NSCLC; Discrete choice experiment (DCE)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort 1: Participants with early stage and advanced/metastatic non-small cell lung cancer (NSCLC)
- Cohort 2: Participants from the general population

SUMMARY:
The purpose of this observational study is to determine participants' preferences for outcomes associated with first-line treatment of advanced/metastatic Non-Small Cell Lung Cancer (NSCLC) using a discrete-choice experiment (DCE).

ELIGIBILITY:
Inclusion Criteria:

The following is the inclusion criteria for pretest interviews and final online survey.

Participants:

* Must be 18 years of age or older
* Must be a US resident.
* Lung cancer participants with a physician diagnosis of NSCLC. Global Perspectives will be involved to suggest alternative strategies to a physician-confirmed diagnosis to ensure that actual cancer participants are recruited.

Exclusion Criteria:

* Not applicable

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study includes pretest interviews with 15 participants diagnosed with non-small cell lung cancer (NSCLC) and 15 participants selected from the general population following the study inclusion criteria. The final survey will be administered online to 150 participants with NSCLC and 500 participants from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Set of relative preference weights for all attribute levels included in the Discrete Choice Experiment (DCE) | At Baseline
Respondents' baseline understanding of attribute descriptions | At Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- RTI Health Solutions, Research Triangle Park, North Carolina, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm